CLINICAL TRIAL: NCT01726673
Title: Effects of Transcranial Direct Current Stimulation Paired With Robotic Arm Therapy on Recovery of Upper Extremity Motor Function in Stroke Patients
Brief Title: Robots Paired With tDCS in Stroke Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Volpe, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-102B
Record Dates: First submitted 2012-10-26; First posted 2012-11-15 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Stroke
Keywords: Stroke; Cerebrovascular Accident; Cerebral Stroke; CVA; Robotic therapy; Upper extremity recovery; tDCS; Non-invasive brain stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS + robotic arm therapy (Experimental): Transcranial Direct Current Stimulation (tDCS) 2mA for 20 minutes over the primary motor cortex (M1) in the affected hemisphere immediately followed by robotic arm therapy for 60 minutes, 3x per week for 12 weeks (36 sessions total)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- tDCS sham + robotic arm therapy (Placebo Comparator): Transcranial Direct Current Stimulation sham condition (0 mA) for 20 minutes over the primary motor cortex (M1) in the affected hemisphere immediately followed by robotic arm therapy for 60 minutes, 3x per week for 12 weeks (36 sessions total)
  Interventions: Device: Placebo sham

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS)
  Other Names: tDCS; Low intensity transcranial DC stimulator; Soterix 1x1
  Arms: tDCS + robotic arm therapy
Device: Placebo sham
  Other Names: tDCS sham
  Arms: tDCS sham + robotic arm therapy

SUMMARY:
The purpose of this study is to evaluate if multiple therapy sessions of Transcranial Direct Current Stimulation (tDCS non-invasive brain stimulation) combined with robotic arm therapy lead to a greater functional recovery in upper limb mobility after stroke than that provided by robotic arm therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* First single focal unilateral lesion with diagnosis verified by brain imaging, which occurred at least 6 months prior
* Cognitive function sufficient enough to understand experiments and follow instructions
* Fugl-Meyer assessment of 7 to 58 out of 66 (neither hemiplegic nor fully recovered motor function in the muscles of the shoulder, elbow, and wrist)

Exclusion Criteria:

* Botox treatment within 6 weeks of enrollment
* Fixed contraction of the affected limb
* Complete flaccid paralysis of the affected limb
* History of hemorrhagic stroke
* Ongoing use of CNS active medications
* Ongoing use of psychoactive medications
* Presence of additional potential tDCS/TMS risk factors including damaged skin at site of stimulation, presence of a magnetically/mechanically active implant, metal in the head, family history of epilepsy, and personal history of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce T Volpe, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States

REFERENCES:
- [Background] Edwards DJ, Krebs HI, Rykman A, Zipse J, Thickbroom GW, Mastaglia FL, Pascual-Leone A, Volpe BT. Raised corticomotor excitability of M1 forearm area following anodal tDCS is sustained during robotic wrist therapy in chronic stroke. Restor Neurol Neurosci. 2009;27(3):199-207. doi: 10.3233/RNN-2009-0470. PMID 19531875
- [Derived] Moretti CB, Hamilton T, Edwards DJ, Peltz AR, Chang JL, Cortes M, Delbe ACB, Volpe BT, Krebs HI. Robotic Kinematic measures of the arm in chronic Stroke: part 2 - strong correlation with clinical outcome measures. Bioelectron Med. 2021 Dec 29;7(1):21. doi: 10.1186/s42234-021-00082-8. PMID 34963502
- [Derived] Moretti CB, Edwards DJ, Hamilton T, Cortes M, Peltz AR, Chang JL, Delbem ACB, Volpe BT, Krebs HI. Robotic Kinematic measures of the arm in chronic Stroke: part 1 - Motor Recovery patterns from tDCS preceding intensive training. Bioelectron Med. 2021 Dec 29;7(1):20. doi: 10.1186/s42234-021-00081-9. PMID 34963501
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized to receive 36 sessions of either active tDCS immediately followed by robotic arm therapy or sham tDCS immediately followed by robotic arm therapy.
Groups:
- tDCS + Robotic Arm Therapy: Transcranial Direct Current Stimulation (tDCS) 2mA for 20 minutes over the primary motor cortex (M1) in the affected hemisphere immediately followed by robotic arm therapy for 60 minutes, 3x per week for 12 weeks (36 sessions total)
  Transcranial Direct Current Stimulation (tDCS)
- tDCS Sham + Robotic Arm Therapy: Transcranial Direct Current Stimulation sham condition (0 mA) for 20 minutes over the primary motor cortex (M1) in the affected hemisphere immediately followed by robotic arm therapy for 60 minutes, 3x per week for 12 weeks (36 sessions total).
  Placebo sham
Period: Overall Study
Arm/Group | tDCS + Robotic Arm Therapy | tDCS Sham + Robotic Arm Therapy
Started | 30 | 24
Completed | 24 | 21
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- tDCS Sham + Robotic Arm Therapy: Transcranial Direct Current Stimulation sham condition (0 mA) for 20 minutes over the primary motor cortex (M1) in the affected hemisphere immediately followed by robotic arm therapy for 60 minutes, 3x per week for 12 weeks (36 sessions total)
  Placebo sham
- Total: Total of all reporting groups
Arm/Group | tDCS + Robotic Arm Therapy | tDCS Sham + Robotic Arm Therapy | Total
Number analyzed (Participants) | 30 | 24 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 30
  >=65 years | 10 | 14 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 19 | 15 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 20 | 13 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Median Change in Upper Extremity Fugl Meyer Assessment Score
Description: The median change in Upper Extremity Fugl-Meyer Score was calculated from baseline to discharge at 12 weeks (immediately following the intervention) and again at 36 weeks (6 months follow-up from the intervention) in each training condition (sham tDCS + robotics arm training vs. active tDCS + robotic arm training). The total Upper Extremity Fugl Meyer score is reported, with a range 0-66 points, and with higher values indicating better functional status.
Time Frame: baseline, discharge at 12 weeks (immediately following the intervention), and follow-up at 36 weeks (6 months after the intervention)
Population: 45 patients completed 36 sessions (3x/week for 12 weeks) of robotic arm training + sham or active tDCS, and 6 month follow-up at 36 weeks. These 45 participants were consequently included in the efficacy analysis.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Groups:
- tDCS + Robotic Arm Therapy: Active Transcranial Direct Current Stimulation (tDCS) 2mA for 20 minutes over the primary motor cortex (M1) in the affected hemisphere immediately followed by robotic arm therapy for 60 minutes, 3x per week for 12 weeks (36 sessions total)
  Transcranial Direct Current Stimulation (tDCS)
Arm/Group | tDCS + Robotic Arm Therapy | tDCS Sham + Robotic Arm Therapy
Number analyzed (Participants) | 24 | 21
scores on a scale
  Median change from baseline to discharge at 12 wks | 4.5 [3 to 8] | 6.0 [4 to 8]
  Median change from baseline to 6 month follow-up | 4 [2 to 7] | 6 [4 to 7.25]
Statistical Analysis 1: Comparison: tDCS + Robotic Arm Therapy vs tDCS Sham + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of median change from baseline to DC immediately following 12 weeks of training was assessed with the upper extremity fugl meyer score in the active vs. sham tDCS conditions. Null hypothesis is that there is no difference in median change in upper extremity fugl meyer score between the active and sham tDCS conditions. A significance level of 0.05 was used (two-tailed); p = 0.256, Mann-Whitney U test — The Mann-Whitney U test was performed to compare median change in upper extremity fugl meyer score from baseline to 12 weeks (discharge) across two separate study conditions (active vs. sham tDCS); U value = 302
Statistical Analysis 2: Comparison: tDCS + Robotic Arm Therapy vs tDCS Sham + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of median change from baseline to week 36 (6 month follow-up) was assessed with upper extremity fugl meyer score for the active vs. sham tDCS conditions. Null hypothesis is that there is no difference in median change in upper extremity fugl meyer score between the active and sham tDCS conditions. A significance level of 0.05 was used (two-tailed); p = 0.222, Mann-Whitney U test — The Mann-Whitney U test was performed to compare median change in upper extremity fugl meyer score from baseline to 36 weeks (follow-up) across two separate study conditions (active vs. sham tDCS); U value = 222

2. Secondary Outcome: Median Change in WOLF Motor Function Test (WMFT)
Description: The median change in performance time for the WOLF motor function test was calculated from baseline to discharge at 12 weeks (immediately following the intervention) and again at 36 weeks (6 months follow-up from the intervention) in each training condition (sham tDCS + robotics arm training vs. active tDCS + robotic arm training). The total WOLF motor function timed score is reported here in seconds, with a range 0-1800 seconds, and with lower values indicating faster completion of task and better functional status.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | tDCS + Robotic Arm Therapy | tDCS Sham + Robotic Arm Therapy
Number analyzed (Participants) | 24 | 21
seconds
  Median change from baseline to discharge at 12 wks | -34 [-235.25 to 0] | -19 [-157 to -1.5]
  Median change from baseline to 6 month follow-up | -103 [-245.5 to -5] | -81.5 [-260.5 to 0]
Statistical Analysis 1: Comparison: tDCS + Robotic Arm Therapy vs tDCS Sham + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of median change from baseline to DC immediately following 12 weeks of training was assessed with the WOLF Motor Function test time score (out of 1800 seconds) in the active vs. sham tDCS conditions. Null hypothesis is that there is no difference in median change in WMFT time score between the active and sham tDCS conditions. A significance level of 0.05 was used (two-tailed); p = 1.0, Mann-Whitney U Test — The Mann-Whitney U test was performed to compare median change in the WMFT time score from baseline to 12 weeks (discharge) across two separate study conditions (active vs. sham tDCS); U Value = 251.5
Statistical Analysis 2: Comparison: tDCS + Robotic Arm Therapy vs tDCS Sham + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of median change from baseline to week 36 (6 month follow-up) was assessed with the WOLF Motor Function test time score (out of 1800 seconds) in the active vs. sham tDCS conditions. Null hypothesis is that there is no difference in median change in WMFT time score between the active and sham tDCS conditions. A significance level of 0.05 was used (two-tailed); p = 0.592, Mann-Whitney U Test — The Mann-Whitney U test was performed to compare median change in the WMFT time score from baseline to 36 weeks ( 6 month follow-up) across two separate study conditions (active vs. sham tDCS); U value = 208.5

3. Secondary Outcome: Median Change in Motor Power Manual Muscle Test Score for the Upper Extremity (MRC)
Description: The median change in Motor Power Manual Muscle Test Score for the upper extremity was calculated from baseline to discharge at 12 weeks (immediately following the intervention) and again at 36 weeks (6 months follow-up from the intervention) in each training condition (sham tDCS + robotics arm training vs. active tDCS + robotic arm training). The total Motor Power Manual Muscle Test Score is reported here, with a range 0-100 points, and with higher values indicating better functional status.
Time Frame: 12 weeks (immediately following the intervention) and 36 weeks (6 months after the intervention)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | tDCS + Robotic Arm Therapy | tDCS Sham + Robotic Arm Therapy
Number analyzed (Participants) | 24 | 21
scores on a scale
  Median change from baseline to discharge at 12 wks | 7 [4 to 9.5] | 7 [5 to 8]
  Median change from baseline to 6 month follow-up | 6 [3 to 11.25] | 6 [4 to 9]
Statistical Analysis 1: Comparison: tDCS + Robotic Arm Therapy vs tDCS Sham + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of median change from baseline to DC immediately following 12 weeks of training was assessed with the Motor Power Manual Muscle Test Score for the upper extremity (out of 100 points) in the active vs. sham tDCS conditions. Null hypothesis is that there is no difference in median change in MRC score between the active and sham tDCS conditions. A significance level of 0.05 was used (two-tailed); p = 0.680, Mann-Whitney U test — The Mann-Whitney U test was performed to compare median change in the MRC score from baseline to 12 weeks (discharge) across two separate study conditions (active vs. sham tDCS); U value = 270.5
Statistical Analysis 2: Comparison: tDCS + Robotic Arm Therapy vs tDCS Sham + Robotic Arm Therapy; Test type: Equivalence — Statistical analysis of median change from baseline to week 36 (6 month FU) was assessed with the Motor Power Manual Muscle Test Score for the upper extremity (out of 100 points) in the active vs. sham tDCS conditions. Null hypothesis is that there is no difference in median change in MRC score between the active and sham tDCS conditions. A significance level of 0.05 was used (two-tailed); p = 0.837, Mann-Whitney U Test — The Mann-Whitney U test was performed to compare median change in the MRC score from baseline to 6 month FU across two separate study conditions (active vs. sham tDCS); U value = 187.5

ADVERSE EVENTS:
Time Frame: Patients were followed for a total of 36 weeks, including the 12 weeks of the study intervention, and the 6 month follow-up period.
Arm/Group | tDCS + Robotic Arm Therapy | tDCS Sham + Robotic Arm Therapy
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/24
Other Adverse Events (participants affected / at risk) | 2/30 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS + Robotic Arm Therapy (N=30) | tDCS Sham + Robotic Arm Therapy (N=24)
Myasthenia Gravis (Nervous system disorders) | 1 (1) | 0 (0) — Subject developed spontaneous eye pstosis at home and was diagnosed with Myasthenia Gravis by treating physician, unrelated to study intervention.
back pain flair up (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject developed flair up of lower back pain as a result of compromised gait pattern after stroke and consequently had to drop out of the study.
seizure (Nervous system disorders) | 0 (0) | 1 (1) — Subject from the sham condition experienced a seizure at home greater than 48 hrs after stimulation, and seizure was determined to be unrelated to study intervention by subject's treating neurologist. Subject was withdrawn from study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT01726673/Prot_SAP_000.pdf